CLINICAL TRIAL: NCT06132295
Title: Adoption of Multiple Strategies to Reduce the Rate of Marker Detachment During Radiotherapy in Patients With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2023-A-037
Record Dates: First submitted 2023-11-07; First posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-07

CONDITIONS: Radiation Therapy; Cancer Patients; Tattooing
MeSH Terms: interventions — Nursing Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nursing care (Experimental): Investigators used in-house-designed radiotherapy red and green light markers to distinguish individual measures after the provision of the initial nursing care to participants, added a homemade health education leaflet to collect data via actual observation, and counted the disappearance or fading of participants' body markers
  Interventions: Other: Nursing care

INTERVENTIONS:
Other: Nursing care — 1. Consistent Schedule for the Replacement of Positioning Line Pens
  2. Tailored Educational Content
  3. Hypoallergenic Adhesive Patches
  4. Enriched Treatment Care Platform
  5. Participants with BMI > 25 and an education level of high school or below, without specific caregivers, were identified by placing a red dot on the treatment record and on the patient's happiness card. Patients with BMI < 25 and an education level of high school or above, with specific caregivers, were identified by placing a green dot on their records.
  6. Individual interventions, educational pamphlets prepared in-house were added, to assess the maintenance status of the positioning marks.

SUMMARY:
Investigators used in-house-designed radiotherapy red and green light markers to distinguish individual measures after the provision of the initial nursing care to participants, added a homemade health education leaflet to collect data via actual observation, and counted the disappearance or fading of participants' body markers

DETAILED DESCRIPTION:
From January 1, 2023 to June 30, 2023, a total of 200 participants were enrolled and undergoing radiation therapy. Inclusion Criteria: clear consciousness who could understand and comprehend Mandarin Chinese. Exclusion Criteria: patients with impaired consciousness or decreased cognitive abilities.

Investigators proposed a set of strategic initiatives :

1. Consistent Schedule for the Replacement of Positioning Line Pens: Consistent Schedule for the Replacement of Positioning Line Pens: Investigators recommend implementing a standardized replacement schedule for positioning line pens, with replacement performed after every 50 uses.
2. Tailored Educational Content: Investigators created personalized educational content tailored to each patient's educational background. This approach ensures that participants can easily understand their treatment plan.
3. Hypoallergenic Adhesive Patches: Investigators offered a variety of hypoallergenic adhesive patches, catering to the skin characteristics of individual participants.
4. Enriched Treatment Care Platform: Investigators commitment extended to creating a comprehensive treatment care platform, which provided guidance on positioning line usage, interactive community features, and practical information.
5. Participants with BMI > 25 and an education level of high school or below, without specific caregivers, were identified by placing a red dot on the treatment record and on the patient's happiness card. Patients with BMI < 25 and an education level of high school or above, with specific caregivers, were identified by placing a green dot on their records.
6. After implementing the red-green light differentiation for radiation therapy and individual interventions, educational pamphlets prepared in-house were added, to assess the maintenance status of the positioning marks.

The number of times the surface marks disappeared or faded during treatment was recorded on the day the participants completed treatment.

ELIGIBILITY:
Inclusion Criteria:

* participants with clear consciousness.
* participants could understand and comprehend Mandarin Chinese.

Exclusion Criteria:

* participants with impaired consciousness or decreased cognitive abilities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
The number of times the surface marks disappeared or faded | The day the participants immediately after the radiotherapy.
  The number of times the surface marks disappeared or faded during treatment was recorded on the day the participants immediately after the radiotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Chung Shan Medical University, Taichung, Taiwan (r.o.c.), Taiwan

IPD SHARING:
Plan to Share IPD: No